CLINICAL TRIAL: NCT04512131
Title: Impact of Dialysis Modality on Coagulation and Platelet Function in Critically Ill Patients: Intermittent Hemodialysis vs. Continuous Renal Replacement Therapy
Brief Title: Impact of Dialysis Modality on Coagulation and Platelet Function
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Associate professor, Seoul National University Hospital
Other Study IDs: Dialysis mode_coagulation
Record Dates: First submitted 2020-08-04; First posted 2020-08-13 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Intermittent hemodialysis: patients who are going to undergo intermittent hemodialysis or patients who are going to switch dialysis mode to intermittent hemodialysis from continuous renal replacement therapy Laboratory test including complete blood count, prothrombin time, activated partial thromboplastin time, protein C, protein S and D-dimer, EXTEM of ROTEM and Multiplate® platelet function analysis will be checked just before dialysis initiation and immediately after dialysis termination
  Interventions: Procedure: dialysis mode
- continuous renal replacement therapy: patients who are going to undergo continuous renal replacement therapy Laboratory test including complete blood count, prothrombin time, activated partial thromboplastin time, protein C, protein S and D-dimer, EXTEM of ROTEM and Multiplate platelet function analysis will be checked within 24 hours after dialysis initiation and 48 hours after taking first blood sample
  Interventions: Procedure: dialysis mode

INTERVENTIONS:
Procedure: dialysis mode — intermittent hemodialysis or continuous renal replacement therapy

SUMMARY:
The investigators will evaluate the impact of dialysis modality (intermittent hemodialysis or continuous renal replacement therapy) in coagulation and platelet function in critically ill patients

DETAILED DESCRIPTION:
An prospective observational study will be conducted to confirm the impact of two dialysis modalitites on coagulation and platelet function in critically ill patients requiring renal replacement therapy using laboratory test, Multiplate and ROTEM.

ELIGIBILITY:
Inclusion Criteria:

• Critically ill adult patients in surgical intensive care unit who require renal replacement therapy

Exclusion Criteria:

* Patients treated with anti-coagulation therapy due to thrombosis/embolism
* Patients who take anti-platelet drug due to cardiac or cerebrovascular diseased
* Patients treated with pharmacological prophylaxis of deep vein thrombosis
* Patients who received blood products within 24 hours of dialysis initiation
* Patients who do not want life-sustaining care including renal replacement therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill adult patients in surgical intensive care unit requiring renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
clotting time (CT) in EXTEM in rotational thromboelastometry (ROTEM) | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of changes in CT in EXTEM of ROTEM (seconds)

SECONDARY OUTCOMES:
Multiplate® platelet function analysis area under curve unit | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of platelet function using Multiplate®
clot formation time (CFT) in EXTEM | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of CFT in EXTEM using ROTEM (seconds)
Amplitude 10 minutes after CT (A10) in EXTEM | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of A10 in EXTEM using ROTEM (mm)
α-angle in EXTEM | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of α-angle in EXTEM using ROTEM (º)
Maximal clot firmness (MCF) in EXTEM | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of MCF in EXTEM using ROTEM (mm)
prothrombin time | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of prothrombin time (seconds)
activated partial thromboplastin time | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of activated partial thromboplastin time (seconds)
Protein C | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of Protein C
Protein S | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of Protein S
fibrinogen | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of fibrinogen
D-dimer | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of D-dimer
platelet count | before and after applying each mode of dialysis (4 hours in intermittent hemodialysis and 48 hours in continuous renal replacement therapy
  the difference of platelet count
the amount of blood transfusion | 24 hours
  the amount of blood transfusion for 24 hours after taking second blood sample
hemodynamic changes | 24 hours
  changes of mean arterial pressure > 20 %, increased vasopressor/inotropics
changes of characteristics or amount of drainage | 24 hours
  changes of characteristics or amount of drainage

OTHER OUTCOMES:
complication related to bleeding | 24 hours
  gastrointestinal bleeding-hematochezia/melena, intra-abdominal bleeding, airway bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT04512131/Prot_SAP_000.pdf